CLINICAL TRIAL: NCT06876558
Title: Exploring the Multimorbidity Burden in Primary Care in Romania
Acronym: MULTIMORB-PC-R
Status: Not yet recruiting | Type: Observational
Sponsor: Internist.Ro (Other)
Collaborators: Transilvania University of Brasov (Other)
Responsible Party: Sponsor
Other Study IDs: A003
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Multimorbidity; General Practice (GP), Primary Care Settings; Specialist Referral
Keywords: multimorbidity; priamary care; specialized care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Primary Care Physicians (PCPs): General practitioners (GPs) actively working in primary care settings. Responsible for managing multimorbid patients in ambulatory settings. Expected proportion: MHalf of the population
- Ambulatory Care Specialists: Specialists involved in outpatient management of chronic diseases (e.g., internal medicine, cardiology, endocrinology).
  Provide secondary care and interact with PCPs in multimorbidity management.

SUMMARY:
Multimorbidity, the coexistence of two or more chronic conditions, is a growing challenge in primary care, significantly impacting healthcare systems worldwide. Its prevalence is rising, particularly among socioeconomically disadvantaged populations, leading to increased healthcare utilization, polypharmacy, and fragmented care. Current clinical guidelines primarily address single-disease management, failing to provide comprehensive strategies for multimorbid patients.

Although multimorbidity has been extensively studied in Western Europe and North America, data on its burden in Romania and other Eastern European countries remain scarce. There is limited knowledge on how primary care physicians (PCPs) in Romania perceive and manage multimorbidity, particularly regarding clinical decision-making, interdisciplinary collaboration, and adherence to treatment guidelines.

This cross-sectional study aims to explore the impact of multimorbidity on Romanian PCPs, assessing their challenges in managing complex patients, their clinical and therapeutic approaches, and their level of comfort with deprescription and guideline adaptation. We will conduct a nationwide survey among primary care physicians and ambulatory specialists to evaluate the prevalence of multimorbidity in their practice, the difficulties they encounter, and potential strategies to improve care delivery.

Key outcomes include the identification of multimorbidity prevalence in ambulatory settings, challenges related to consultation time and treatment complexity, barriers to interdisciplinary collaboration, and the balance between defensive and proactive medicine. Findings will provide valuable insights to guide policy changes, enhance clinical training, and promote patient-centered approaches in primary care

DETAILED DESCRIPTION:
Background and Rationale Multimorbidity, defined as the presence of two or more chronic conditions in the same individual, is a growing concern in global healthcare. It significantly impacts healthcare systems, increasing hospital admissions, prolonging hospital stays, and elevating healthcare costs. In the European Union, it is estimated that at least 50 million people suffer from multimorbidity, and this number is expected to rise with aging populations (Rijken et al., 2013).

Patients with multimorbidity experience worse health outcomes compared to those with a single chronic disease, including higher mortality rates, reduced functional capacity, lower health-related quality of life (HRQoL), and a greater prevalence of depression (Menotti et al., 2001, Christine Vogeli et al., 2007). Managing multimorbidity is particularly complex due to polypharmacy and the risk of adverse drug interactions. The current disease-specific clinical guidelines, which primarily focus on single-disease management, often fail to address the multifaceted needs of multimorbid patients (Kristen Anderson et al., 2017).

State of the Art Multimorbidity research has been widely conducted in high-income Western European countries and North America, leading to established frameworks for care models, clinical guidelines, and integrated management strategies. However, research on multimorbidity in Eastern European healthcare systems remains scarce. Romania, in particular, lacks comprehensive data on multimorbidity prevalence, its impact on primary care, and physicians' perspectives on its management.

In many healthcare systems, general practitioners (GPs) are at the frontline of multimorbidity management, yet they face substantial challenges, including limited consultation time, scarce resources, and difficulties in coordinating with specialists. Multimorbid patients require personalized care plans, often leading to guideline deviations that may cause physician anxiety about potential medical and legal repercussions. Understanding how Romanian primary care physicians navigate these challenges is essential to improving patient outcomes and optimizing healthcare delivery.

Knowledge Gap

Despite the increasing prevalence of multimorbidity in Romania, there is little empirical evidence regarding:

The proportion of multimorbid patients seen in primary care. The specific challenges physicians face in managing these patients. The role of interdisciplinary collaboration and the barriers to integrated care.

The balance between defensive medicine and proactive deprescription strategies. The impact of multimorbidity on physicians' clinical decision-making and their adherence to single-disease guidelines.

By addressing these gaps, this study aims to provide valuable insights into how multimorbidity affects clinical practice in Romania and identify potential improvements in patient-centered care.

Objectives

This study aims to explore the impact of multimorbidity on primary care physicians in Romania, focusing on:

The prevalence of multimorbidity in ambulatory care. The challenges faced by GPs, including time constraints, polypharmacy, and resource limitations.

Difficulties in interdisciplinary collaboration and care coordination. The use of defensive vs. proactive medicine in multimorbidity management. The influence of multimorbidity on adherence to clinical guidelines and physician decision-making.

Potential solutions to improve multimorbidity management, including extending consultation times, enhancing interdisciplinary collaboration, and integrating multimorbidity-focused guidelines into primary care.

Methods Study Design This is a cross-sectional survey-based study conducted among primary care physicians and ambulatory care specialists in Romania. The survey will assess multimorbidity's impact on clinical decision-making, patient management strategies, and interdisciplinary collaboration. A semi-qualitative component will be included to gather in-depth insights from physicians.

Study Population

Inclusion Criteria:

Active medical practice in Romania. Experience in managing patients with multimorbidity. Willingness to participate in the study. Exclusion Criteria: None. Data Collection Survey Distribution: The survey will be disseminated electronically and in print among primary care physicians in Romania and the Balkan region.

Survey Components:

Demographic information: Age, gender, years of experience, practice setting. Clinical workload: Average number of patients seen per day, proportion of multimorbid patients.

Management strategies: Approaches to polypharmacy, deprescription practices, time allocation for multimorbid patients.

Physician perceptions: Challenges faced, levels of comfort with guideline deviations, attitudes toward interdisciplinary collaboration.

Data Processing and Analysis: Quantitative data will be analyzed using descriptive statistics, while qualitative responses will be thematically analyzed.

Outcome Measures

Primary Outcomes:

Proportion of multimorbidity, single morbidity, and non-comorbid patients in ambulatory care.

Identification of challenges related to consultation time, treatment complexity, and polypharmacy.

Assessment of preventive strategies (smoking cessation, alcohol reduction, diet, physical activity, sleep, and social engagement).

Secondary Outcomes:

Barriers to interdisciplinary collaboration and care coordination. Patterns of defensive medicine versus active deprescription practices. Levels of physician anxiety related to adherence to clinical guidelines. Expected Impact

This study will provide evidence on the prevalence and impact of multimorbidity in Romanian primary care. It aims to inform policymakers, healthcare administrators, and medical educators on how to improve multimorbidity management through:

Better allocation of resources and consultation time. Training programs focused on multimorbidity care strategies. Development of integrated care pathways that support interdisciplinary collaboration.

By addressing the challenges faced by primary care physicians, this study will contribute to a more effective and patient-centered approach to multimorbidity management in Romania

ELIGIBILITY:
Inclusion Criteria:

* Active AMBULATORY CARE medical practice in Romania.
* Experience in managing patients with multimorbidity.
* Willingness to participate in the study.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of primary care physicians (PCPs) and ambulatory care specialists actively working in Romania. Participants will be recruited from urban and rural primary care clinics, outpatient specialist practices, and ambulatory care centers across various regions of the country. The survey will be distributed through national and local medical associations, professional networks.
  The expected prevalence of multimorbidity is estimated at 20%. This requires a minimum of 246 completed surveys to achieve a 95% confidence level with a 5% margin of error.
  This population will represent a diverse group of healthcare professionals who are directly involved in the management of multimorbid patients in outpatient settings, ensuring a comprehensive understanding of the challenges and strategies associated with multimorbidity care in Romania.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of multimorbidity | baseline
  Prevalence of multimorbidity in primary care (percentage of patients)
Proportion of single morbidity | baseline
  Proportion of single morbidity (percentage) in primary care practice
Proportion of non comorbid patients | Baseline
  Proportion percentage out of total) of non comorbid patients in primary care versus specialized ambulatory care according to specialty.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea NECULAU, MD, Study Chair — Universitatea Transilvania Brasov; Silvia Sovaila, MD, Principal Investigator — Universitatea Transilvania Brasov; Adrian PURCAREA, MD, Study Director — Internist.Ro
Locations (1):
- Universitatea Transilvania Brasov School of Medicine, Brasov, Romania

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: April 2025-April 2030
Access Criteria: Eligibility for Data Access:
  Data will be shared with qualified researchers affiliated with academic institutions, healthcare organizations, or research institutions conducting studies related to multimorbidity, primary care, or health services research.
  The request must specify the intended scientific objectives, planned statistical analyses, and potential contributions to the field.
  Proposals must align with ethical and legal standards for data privacy and patient confidentiality.
  Data Sharing Mechanism:
  Researchers must submit a formal request detailing their proposed analyses, methodologies, and intended outcomes.
  Requests can be submitted via email to the study sponsor or principal investigator, along with the necessary documentation.

REFERENCES:
- [Background] Rijken,M. and Struckmann,V. and Dyakova,M. and Melchiorre, M. G. and Rissanen,S. and Ginneken,E. van, 20133386107, English, Journal article, Belgium, 1356-1030, 19, (3), Brussels, Eurohealth, (29-31), European Observatory on Health Systems and Policies, ICARE4EU: improving care for people with multiple chronic conditions in Europe., (2013)
- [Background] Anderson K, Foster M, Freeman C, Luetsch K, Scott I. Negotiating "Unmeasurable Harm and Benefit": Perspectives of General Practitioners and Consultant Pharmacists on Deprescribing in the Primary Care Setting. Qual Health Res. 2017 Nov;27(13):1936-1947. doi: 10.1177/1049732316687732. Epub 2017 Jan 12. PMID 29088989
- [Background] Menotti A, Mulder I, Nissinen A, Giampaoli S, Feskens EJ, Kromhout D. Prevalence of morbidity and multimorbidity in elderly male populations and their impact on 10-year all-cause mortality: The FINE study (Finland, Italy, Netherlands, Elderly). J Clin Epidemiol. 2001 Jul;54(7):680-6. doi: 10.1016/s0895-4356(00)00368-1. PMID 11438408